CLINICAL TRIAL: NCT00936442
Title: ARimidex Therapy Compliance Electronic MonitorIng System. A Study to Evaluate the Impact of Educational Material on the Adherence to Treatment With Adjuvant Anastrozole for Postmenopausal Women With Hormone Sensitive Early Breast Cancer
Brief Title: Arimidex Therapy Compliance Electronic Monitoring System
Acronym: ARTEMIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Aardex Pharmionic (Industry)
Responsible Party: Sponsor
Other Study IDs: D5390L00076
Record Dates: First submitted 2009-07-06; First posted 2009-07-10 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Compliance; Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance | interventions — Anastrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Standard treatment: 12-month follow-up of anastrozole treatment according to SmPC and current clinical practice.
  Interventions: Drug: Anastrozole
- Group B: Standard treatment + educational material: 12-month follow-up of anastrozole treatment according to SmPC and current clinical practice plus reception of educational material on regular basis.
  Interventions: Drug: Anastrozole; Other: Educational materials

INTERVENTIONS:
Drug: Anastrozole — (Standard Treatment) 12-month follow-up of anastrozole treatment according to SmPC and current clinical practice.
Other: Educational materials — Reception of educational material on regular basis.
  Groups: Group B

SUMMARY:
ARTEMIS is a study to assess how educational material affects overall adherence to anastrozole by evaluation of patients' electronically compiled dosing histories. Patients' dosing times are compiled electronically using Medication Event Monitoring System" (MEMS®) in order to be able to gather accurate, objective and up-to-date patients' dosing histories. For subjects in Group A, the control group, the adherence to anastrozole in the standard clinical practice will be evaluated. For subjects in Group B, on top of the standard clinical practice, they will also receive educational material by mail at week 0 (study registration), week 2, week 4, week 6, week 8, week 12, month 5, month 7, and at month 10. This procedure is the same as in the ongoing CARIATIDE study. One of the reasons of poor adherence (either early discontinuation of the treatment or missing doses while still engaged to the therapy) can be some side effects experienced by the patients during the anastrozole treatment. Recording the reasons at discontinuation allows us to identify reasons for treatment discontinuation. Recording reasons of anastrozole interruptions during the study period allows us to relate these events to patients' adherence to anastrozole. During the study, no pro-active safety data collection will take place. Spontaneous reported adverse drug reactions (ADRs) will be reported according to local post-marketing pharmacovigilance regulations.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with hormone sensitive early breast cancer.
* Documented decision of treatment with anastrozole which will start in 13 weeks according to current SmPC OR current treatment with anastrozole according to current SmPC, that has not exceeded thirteen weeks before enrollment.
* Subjects who accept to use MEMS® monitors to automatically compile their drug dosing histories.

Exclusion Criteria:

* Concomitant or previous use of adjuvant tamoxifen, letrozole or exemestane for the current tumour.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff or staff at the study site).
* Participation in another clinical study with an investigational product during the last 3 months.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal women with hormone sensitive early breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall adherence to anastrozole | 2/year (after 6 months and after one year)

SECONDARY OUTCOMES:
Patients' persistence with anastrozole | 2/year (after 6 months and after one year)
Execution of the dosing regimen | 2/year (after 6 months and after one year)
Reasons for treatment discontinuation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Nogaret, Principal Investigator — Jules Bordet Institute
Locations (4):
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Overpelt